CLINICAL TRIAL: NCT03674632
Title: Mother-infant Signalling During Lactation Following Late Preterm and Early Term Delivery: An Investigation of Physiological, Psychological and Anthropological Factors
Brief Title: Breastfeed a Better Youngster: the BABY Study
Acronym: BABY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University College, London (Other)
Collaborators: Beijing Children's Hospital (Other)
Responsible Party: Principal Investigator, Mary Fewtrell, Professor in pediatric nutrition, University College, London
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 18PE15
Record Dates: First submitted 2018-08-29; First posted 2018-09-17 (Actual); Last update posted 2020-11-04 (Actual); Status verified 2020-11

CONDITIONS: Breastfeeding; Breastfeeding, Exclusive; Infant Behavior; Psychological Stress; Breast Milk Expression; Infant Development
Keywords: breastfeeding; maternal stress; infant behavior; infant development; relaxation
MeSH Terms: conditions — Breast Feeding; Infant Behavior; Stress, Psychological; Breast Milk Expression

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- relaxation meditation tape (Experimental): Participants in this arm will be asked to use the relaxation therapy during the feed at least once a day. Participants will be given a diary to record when it is used. Participants will be encouraged to use the tape as often as they find it helpful.
  Interventions: Behavioral: Relaxation meditation tape
- Normal care (No Intervention): Participants in this arm will receive normal care from the Beijing Children Hospital

INTERVENTIONS:
Behavioral: Relaxation meditation tape — The tape used in this study is based on a meditation CD designed for breastfeeding mother (Menelli, 2004). The recording will be transcribed and translated into Chinese language by a certified yoga therapist.
  Arms: relaxation meditation tape

SUMMARY:
This research will investigate different aspects of the 'signalling' between mother and infant during breastfeeding in a stressful situation following late preterm and early term delivery, when breastfeeding is often challenging. The researcher will conduct a single-blinded randomised controlled trial in Chinese mothers who deliver a late preterm infant (LPI; 34 0/7-36 6/7 weeks of gestation) and mothers who deliver a early term infant (ETI; 37 0/7-37 6/7) and plan to exclusively breast-feed.This study will investigate the role of the milk and infant gut microbiome as a potential 'signal' in this process. A relaxation intervention (meditation tape) will be used to reduce stress levels in mothers who are expressing breast-milk or breastfeeding their infant (born at 34 0/7-37 6/7 weeks completed gestation). This study will investigate whether lower levels of stress in the mother result in more successful and effective breastfeeding, leading to improved infant outcomes (better growth, longer sleep duration and reduced crying).

DETAILED DESCRIPTION:
Participants will be recruited while they are in the maternity hospital. A baseline assessment will be conducted during the 1-week postpartum home visit, with another study visit at 8 weeks after delivery. After obtaining written informed consent, subjects will be randomly assigned to either the intervention arm or control conditions (standard management). Participants will be told that the aim of the study is to investigate factors that may make breastfeeding easier for mothers with a LPI and ETI, so they can breast-feed for longer. They will not be told about the randomisation until the end of the study, as this knowledge would most likely lead to mothers in the control group using some form of relaxation therapy. Background characteristics of mothers and their early feeding experiences will be recorded.

Participants can choose to complete the questionnaires on paper or online in their own time after the study visit. A breast milk sample will be collected pre-feed and infant anthropometry will be assessed by a trained nurse pre-feed at each home visit. Feed duration will be noted by the trained nurse. Stool samples of infants who were born vaginally will be collected by a trained nurse at baseline and at 8-weeks. At 3-month and 6-month postpartum, there will be a telephone contact to the participants for follow-up. Participants will be invited to complete the infant questionnaires again on paper or online in their own time.

ELIGIBILITY:
Inclusion Criteria:

* Primiparous mother with singleton pregnancy who is breastfeeding her late preterm infants
* Infant is singleton born at 34 0/7-37 6/7 weeks of gestation.
* Mother and infant are generally healthy (free of serious diseases that can affect breastfeeding or nursing infant, or energy balance of the infant).
* No current involvement in other research studies that can potentially affect any of outcome measures.

Exclusion Criteria:

* Infant with serious underlying or chronic disease*
* Mothers who smoke
* Infant receiving any medication regularly

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 96 (Actual)
Dates: Start 2018-11-25 (Actual); Primary Completion 2020-10-31 (Actual); Study Completion 2020-10-31 (Actual)

PRIMARY OUTCOMES:
Changes in maternal stress from baseline to 8 weeks postpartum | 8 weeks
  Measurement for maternal stress will use the Cohen's Perceived Stress Scale (PSS). The PSS is a 14-item psychological self-rating scale for measuring the perception of stress on a scale of five, from 0 (never) to 4 (very often).

SECONDARY OUTCOMES:
Infant weight | 8 weeks
  Infant weight will be measured at baseline and the 8-week home visit (unit kg)
Infant length | 8 weeks
  Infant length will be measured at baseline and the 8-week home visit (unit cm)
Infant head circumference | 8 weeks
  Infant head circumference will be measured at baseline and the 8-week home visit (unit cm)
Infant temperament | 8 weeks
  Measured using the revised Rothbart Infant Behaviour Questionnaire (RIBQ) at 2 months of age. The RIBQ is a 7-point Likert scale, from 1 (never) to 7 (always). Three major dimensions will be used for the assessment of infant temperament; surgency/extraversion, negative affectivity and orienting/regulation.
Infant behaviour | 8 weeks
  Measured by 3-day infant behaviour diary (average mins per day spent in each behavioural state). The diary consists of a time scale for 72 hours, which is divided into 15 minutes segments, and has five categories of behaviour: Sleeping, Awake and content, Fussy, Crying and Feeding.
Infant appetite | 8 weeks
  Measured using the Baby Eating Behaviour Questionnaire (BEBQ) at 2 months of age. It consists of 18 items designed to measure four traits: "enjoyment of food" (4 items), "food responsiveness" (5 items), "slowness in eating" (4 items), and satiety responsiveness" (5 items). The mothers in this study will be asked to rate all items based on a scale from 1 (never) to 5 (always).
Composition of milk macronutrients (fat, protein, carbohydrate） | 10 minutes
  Measured by Mid-infrared milk analyser (unit is g/100ml)
Composition of microbiota in breastmilk samples at one week and 8-week postpartum | 8 weeks
  Measured using the 16S rRNA based amplicon sequencing technique
Composition of microbiota in stool samples at one week and 8-week postpartum | 8 weeks
  Measured using the 16S rRNA based amplicon sequencing technique
Breast milk volume at 8 weeks | 8 weeks
  The milk volume will be measured using the test-weighing method.
Energy content of the milk | 10 minutes
  The energy content will estimated from the milk volume measurement provided by Mid-infrared milk analyser in ml and kcal/100ml

CONTACTS AND LOCATIONS:
Overall Officials: Mary Fewtrell, PhD, Principal Investigator — University College, London
Locations (2):
- China (2):
  - Beijing Children Hospital, Beijing
  - Zhuang Wei, Beijing

IPD SHARING:
Plan to Share IPD: No
The IPD will only be used in a PhD thesis and further investigations

REFERENCES:
- [Derived] Yu J, Wells J, Wei Z, Fewtrell M. Effects of relaxation therapy on maternal psychological state, infant growth and gut microbiome: protocol for a randomised controlled trial investigating mother-infant signalling during lactation following late preterm and early term delivery. Int Breastfeed J. 2019 Dec 16;14:50. doi: 10.1186/s13006-019-0246-5. eCollection 2019. PMID 31889973